CLINICAL TRIAL: NCT05081336
Title: Low-density Lipoprotein Cholesterol Reduction With State-of-the-art Therapy in Secondary Prevention and Major Cardiovascular Adverse Events: Republic of Srpska Registry
Acronym: RS-ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Clinical Centre of Republic of Srpska (Other)
Responsible Party: Principal Investigator, Bojan Stanetic, Assistant Prof. Bojan Stanetic, MD, PhD, University Clinical Centre of Republic of Srpska
Other Study IDs: 022021
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Acute Coronary Syndrome; Dyslipidemias
MeSH Terms: conditions — Acute Coronary Syndrome; Dyslipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; alirocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High-intensity statin
  Interventions: Drug: Statin
- High-intensity statin plus ezetimib
  Interventions: Drug: Statin
- High-intensity statin plus ezetimib plus PCSK9 inhibitor
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Statin — Statin +/- ezetimib +/- Alirocumab
  Other Names: Ezetimib; Alirocumab

SUMMARY:
Recent trials have demonstrated that a reduction in low-density lipoprotein cholesterol (LDL-C) reduces cardiovascular adverse events following acute coronary syndrome (ACS). However, the data coming from the real-world setting are limited. Therefore, the aim of the study is to assess the association between LDL-C changes with prognosis in patients who survive ACS.

Patients with ACS will be followed for mortality and major events for at least 1 year. Changes in LDL-C between the ACS and a 6- to 10-week follow-up visit will be analysed. The associations between quartiles of LDL-C change and therapy intensity with outcomes will be investigated using adjusted Cox regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presented with acute coronary syndrome in one of hospitals in Republic of Srpska
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Major Cardiovascular Adverse Events | 1 year
  All-cause death, Acute Coronary Syndrom, Need for Myocardial Revascularization

SECONDARY OUTCOMES:
LDL reduction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bojan M Stanetic, MD, PhD, Principal Investigator — University Clinical Centre of the Republic of Srpska
Locations (1):
- University Clinical Centre of the Republic of Srpska, Banja Luka, Republika Srpska, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code